CLINICAL TRIAL: NCT02161978
Title: Micro and Macro Vascular Dysfunction Induced by Antiangiogenic Therapy: Identification of New Vascular Biomarkers (DYVA-AAGG)
Brief Title: Vascular Dysfunction and Antiangiogenic Therapy
Acronym: DYVA-AAGG
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2011-A00441-40
Record Dates: First submitted 2014-06-02; First posted 2014-06-12 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Solid Tumor; Tumor Angiogenesis; Endothelial Dysfunction; CML (Chronic Myelogenous Leukemia)
Keywords: antiangiogenic; cancer; vascular; biomarker; tyrosine kinase inhibitor
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
project is a pilot prospective, longitudinal, before-after, open label multicentric study.

DETAILED DESCRIPTION:
Antiangiogenic drugs and tyrosine kinase inhibitor (TKI) represent a new therapeutic issue in the treatment of several neoplasic tumors (colon, kidney, breast, lung, skin) and hemopathy. Antiangiogenic drugs acts through neutralization of the activity (e.g. bevacizumab) or the inhibition of post-receptor tyrosine kinase pathways (e.g. sunatinib, sorafenib), leading to a reduction and inhibition of the tumoral tissular neovascularization. Due to the ubiquitous role of and the systemic administration of the antiangiogenic drugs, almost all of them are responsible for several side effects, many involving the cardiovascular system (e.g. arterial hypertension, cardiomyopathies, proteinuria, bleedings,...) and leading to a reduction of the doses or withdrawal of the treatment. To date, the mechanism and the impact of these cardiovascular effects is not well understood involving structural (i.e. capillary rarefaction) and functional vascular dysfunction (i.e. vasomotor dysfunction, stiffening).

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 years old treated for a solid tumor (kidney, pancreas, breast, lungs, skin) with line antiangiogneic therapy and hemopathy
* Antiangiogneic therapy can be: bevacizumab, anti- (e.g. sunitinib, sorafenib), proteinate kinases inhibitor (e.g.temsirolimus ) or everolimus or any new allowed therapy with expected antiangiogenic properties and tyrosine kinase inhibitor.
* Expected life span > 6 months
* Clinical state allowing investigations
* A blood glucose and lipid tests within the last 3 months

Exclusion Criteria:

* Informed consent not obtained
* Patients presenting a clinical state which does not allow for the performance of the vascular investigations (agitation, cutaneous wound, major asthenia, acute dyspnoea, cadiac arhythmia)
* Pregnant women
* Patients > 18 yrs old protected by the french law
* Patients without national health insurance
* Patients included in another biomedical study (this criteria is relative to the other studies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for a solid tumor (kidney, pancreas, intestinal, breast, lungs, skin) requiring a first or second line antiangiogenic therapy and Hemopathy
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2012-02-09 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Changes induced by antiangiogenic drugs and tyrosine kinase inhibitor in the vascular ultrasound variables | 24 months
  arterial stiffness, diameter and resistance will be performed using echotracking technologies.

CONTACTS AND LOCATIONS:
Overall Officials: Samir HENNI, MD, Principal Investigator — University hospital, Angers, FRANCE
Locations (1):
- University Hospital Angers, Angers, France